CLINICAL TRIAL: NCT06672614
Title: Effect of Five Days of Postexercise Hot-Water Immersion on Exercise Performance in Hypoxia
Brief Title: Postexercise Hot-Water Immersion on Exercise Performance in Hypoxia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nipissing University (Other)
Responsible Party: Principal Investigator, Geoff Hartley, Associate Professor, Nipissing University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NUREB # 103807
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Heat Exposure; Exercise Training
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Masking Description: Considering that the hot water immersion protocol will be easily perceptible to the participants, it will not be possible to blind them from their group assignment. Also, the investigators will be required to set the water temperature for the immersion protocol following each exercise session, so they will also be aware of group assignments during the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-Exercise Hot Water Immersion (Experimental): Participants will cycle for 60 minutes at 50% of maximal oxygen uptake (VO2 max) followed by 30 minutes post-exercise hot water immersion (40oC) for 5 consecutive days.
  Interventions: Other: Post-Exercise Hot Water Immersion
- Control group (Active Comparator): Participants will cycle for 60 minutes at 50% of maximal oxygen uptake (VO2 max); however, there will be not water immersion following exercise.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Post-Exercise Hot Water Immersion — Participants will cycle for 60 minutes at 50% of maximal oxygen uptake (VO2 max) followed by 30 minutes post-exercise hot water immersion (40oC) for 5 consecutive days.
  Arms: Post-Exercise Hot Water Immersion
Other: Control Group — Participants will cycle for 60 minutes at 50% maximal oxygen uptake (VO2 max) for 5 consecutive days. There is no water immersion following the exercise.
  Arms: Control group

SUMMARY:
The purpose of this study is to determine the effect of 5 days post-exercise hot water immersion on exercise performance at simulated altitude.

DETAILED DESCRIPTION:
Human performance is compromised at altitude due to a lower partial pressure of oxygen and subsequent reductions in the convective transport of oxygen to tissue. Long-term acclimation to attitude incurs physiological adaptations that result in a near return to sea-level performance; however, the time required (~2 weeks) for such adaptations is often logistically challenging for athletes, military personnel or other individuals who reside at sea level. Recent research suggests that physiological acclimation to heat stress (i.e., heat acclimation) and altitude (i.e., hypoxia) share similar cellular adaptations, namely an up-regulation of Hypoxia-inducible factor 1 (HIF-1) and various heat shock proteins. Therefore, it is hypothesized that heat acclimation may provide physiological protection from reduced oxygen transport to the tissue and enhance performance at altitude. This cross-tolerance model is supported by traditional heat acclimation protocols (i.e., submaximal exercise in hot ambient temperature); however, it has not been tested with passive exposure to heat stress through post-exercise hot water immersion.

ELIGIBILITY:
Inclusion Criteria:

* Physically active (minimum of 90 minutes of moderate-intensity exercise per week)

Exclusion Criteria:

* Cardiovascular disease
* resident of >1500 m above sea-level in the past year;
* history of fainting

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Time-Trial Performance in hypoxia conditions | 30 minutes
  Results of a 16 km time-trial test conducted at an fraction of inspired oxygen (FiO2) of 0.14

SECONDARY OUTCOMES:
Pulse oxygen saturation during exercise | 30 minutes
  Capillary oxygen saturation measured on the earlobe throughout the time-trial tests using pulse oximetry.
Skin temperature during exercise | 90 minutes
  Skin temperature measured throughout the time trial-tests and exercise training intervention using temperature probes attached to the calf, thigh, chest and arm, from which weighted averages are calculated.
Core temperature during exercise | 90 minutes
  Core body temperature measured throughout the time-trial tests and exercise training interventions using a rectal temperature probe.
Heart Rate during exercise | 90 minutes
  Heart rate will be measured throughout the time trial tests and exercise training interventions using a wireless (Polar) heart rate chest strap.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey L Hartley, PhD, Principal Investigator — Nipissing University
Locations (1):
- Nipissing University, North Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the study, after de-identification, will be made publicly available using an online data repository.
Supporting Information: SAP, Analytic Code
Time Frame: Data will be made available immediately following publication with no end date.
Access Criteria: Any purpose.